CLINICAL TRIAL: NCT04504513
Title: Expanded Access Program: Trilaciclib for Chemotherapy-induced Myelosuppression in Patients Receiving Chemotherapy for Small Cell Lung Cancer
Brief Title: Expanded Access to Trilaciclib for Patients Receiving Chemotherapy for Small Cell Lung Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: G1 Therapeutics, Inc. (Industry)
Collaborators: Bionical Emas (Industry)
Responsible Party: Sponsor
Other Study IDs: G1T28-501
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Myelosuppression Adult; Chemotherapeutic Toxicity; Small Cell Lung Cancer
Keywords: Lung Cancer; Small Cell Lung Carcinoma; Small Cell Lung Cancer Extensive Stage; Small Cell Lung Cancer Limited Stage; Small Cell Lung Cancer Metastatic; Chemotherapy-induced Neutropenia; Chemotherapy-induced Anemia; CDK 4/6 Inhibitor; trilaciclib; etoposide; carboplatin; cisplatin; topotecan; checkpoint inhibitor; myelosuppression; cyclin-dependent kinase 4/6 inhibitor; myelopreservation; Real World Data; chemotherapy-induced myelosuppression
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — trilaciclib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib is a highly potent, selective, and reversible cyclin-dependent kinase 4/6 inhibitor administered intravenously prior to chemotherapy for chemotherapy-induced myelosuppression (CIM).
  In patients being treated for SCLC, trilaciclib transiently maintains G1 cell cycle arrest of hematopoietic stem and progenitor cells (HSPCs) in the bone marrow, thus protecting the cells from damage by cytotoxic chemotherapy (myelopreservation). This can reduce chemotherapy-related toxicity, making chemotherapy safer and more tolerable, and also reduce the need for rescue interventions that address the effects of myelosuppression, such as growth factors or blood and platelet transfusions.
  Other Names: G1T28

SUMMARY:
The purpose of this expanded access protocol is to provide access to trilaciclib for chemotherapy-induced myelosuppression in patients receiving chemotherapy as a treatment for small cell lung cancer (SCLC).

Patients will receive trilaciclib intravenously as a 30-minute infusion prior to chemotherapy dosing and on each day that chemotherapy is administered.

Supplementary to providing access to trilaciclib, this expanded access program will also capture Real World Data to help inform subsequent trilaciclib development.

Requests for access to trilaciclib will be managed by Bionical Emas. G1 Therapeutics will review eligibility of, as well as complete a medical review of, each patient access request.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require treatment with either intravenous etoposide + platinum (carboplatin or cisplatin) ± an anti-PDL1 or anti-PD1 checkpoint inhibitor OR intravenous topotecan
* Pathologically confirmed diagnosis of SCLC
* Extensive-stage or limited-stage SCLC; patients with limited-stage SCLC receiving chemotherapy with concurrent radiation are NOT eligible.
* Age ≥ 18 years
* ECOG 0 to 2
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L at time of initiation of therapy in this EAP
* Platelet count ≥ 100 x 10^9/L at time of initiation of therapy in this EAP
* Glomerular filtration rate (GFR) of ≥ 20 mL/minute at time of initiation of therapy in this EAP
* Total bilirubin ≤ 1.5x ULN (upper limit normal) at time of initiation of therapy in this EAP
* AST or ALT ≤ 2.5x ULN (≤ 5x ULN in the presence of liver metastases) at time of initiation of therapy in this EAP
* QTcF interval ≤ 450 msec (males) or ≤ 470 msec (females) at screening (confirmed on repeat). For patients with ventricular pacemakers, QTcF ≤ 500 msec
* No personal or family history of long QT syndrome
* Female patient is not lactating or currently pregnant, or plans to become pregnant, while participating in this expanded access program
* Female patients of reproductive potential agree to use effective contraception while in the program and for at least 3 weeks after the last dose of trilaciclib
* Patient agrees not to participate in another expanded access program or clinical trial with an experimental treatment during participation in this EAP
* Active clinical trial with trilaciclib is not available (or if available, it is not appropriate) for the patient

Exclusion Criteria:

* Patients requiring treatment with oral etoposide or oral topotecan
* Patients outside of the United States

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: G1 Therapeutics policy on expanded access — https://www.g1therapeutics.com/patients/access-to-investigational-therapies/